CLINICAL TRIAL: NCT06519461
Title: Effects of a Family-centered Teaching Model on Intern's Perceptions and Children's Occupational Performance
Brief Title: A Family-centered Teaching Model in Pediatric Occupational Therapy Internship
Acronym: FACTmodel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jung-Jiun Shie (Other)
Responsible Party: Sponsor-Investigator, Jung-Jiun Shie, assistant professor, National Pingtung University
Organization: National Pingtung University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MOST108-2637-H-471-001
Record Dates: First submitted 2024-07-13; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Internship and Residency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- family-centered teaching model group (Experimental): The family-centered teaching group provided knowledge and skills of family-centered services for interns in internship
  Interventions: Behavioral: Family-centered teaching model
- conventional family approach group (No Intervention): The conventional family approach provided interns to interact with children in internships.

INTERVENTIONS:
Behavioral: Family-centered teaching model — The program comprised two parts: (1) Didactic lessons: and (2) Hands-on practice. The didactic lessons were designed to prepare interns' knowledge and skills. The hands-on practice were designed to provide opportunities of family-centered experience to work with caregivers and children.
  Arms: family-centered teaching model group

SUMMARY:
Most of the occupational therapy students received the knowledge of family-centered services when they studies in universities, however, the experience of family-centered practice during internships is limited. The purpose is to design a family-centered teaching model and to examine the effects of the teaching model. The positive results showed on students' perceptions and children's occupational performance.

DETAILED DESCRIPTION:
The study examined the differences of interns' perceptions of services toward family-centeredness and children' occupational performance between a family-centered teaching (FACT) model and a conventional family approach incorporated in internships. A two-group quasi-experimental design was employed. Participants included 49 interns, 44 caregivers, and 45 children with disabilities under six-year-old. The perceptions of interns toward FCS in both groups were measured using the Chinese version of the "Measure of Processes of Care-Service Provider" (C-MPOC-SP) at the pre- and post- tests. Children' occupational performance in both groups was rated using the "Canadian Occupational Performance Measure" (COPM) for the pre- and post-tests. Interns in the experimental group demonstrated a significant increase in two of the four C-MPOC-SP subscales compared to their counterparts. Children' scores improved significantly in COPM performance subtest for experimental group, but not on the COPM satisfaction subscale.

ELIGIBILITY:
Inclusion Criteria:

1. Children with developmental delays/disabilities and their caregivers
2. Children with developmental delays/disabilities under six years old
3. The caregivers of the children with disabilities are aged 20 years old or older
4. The caregivers of the children with disabilities or delays can follow the instruction to administer the assessment
5. Students are participating in internships of the pediatric occupational therapy clinical unit at the hospitals.

Exclusion Criteria:

* Caregiver suffered from mental illness and had difficulty to complet the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2021-10-16 (Actual); Study Completion 2021-10-16 (Actual)

PRIMARY OUTCOMES:
The 49 interns' family-centered behaviors including four types of behaviors were measured by the self-reported questionnaire of "Measure of Processes of Care for Service Providers" | at the beginning and the end of the internship; an average of 12 weeks
  The "Measure of Processess of Care-Service Provider" can measure four types of famly-centered behaviors such as (1) Showing Interpersonal Sensitivity; (2) Providing General Information; (3) Communicating Specific Information; (4) Treating People Respectfully. The questionnire is a reliable and valid self-reported questionnaire The questionnaire comprises 27 items in which each item has a 7-point Likert scale from 1 (not at all) to 7 (to a very great extent).
The performance and satisfaction scales of occupational performance for 45 children in both groups were assessed by a semi-structured interview questionnaire of "Canadian Occupational Performance Measure" reported by their caregivers. | at the beginning and the end of the internship; an average of 12 weeks
  The occupational performance assessed by the "Canadian Occupational Performance Measure" includes the performance on the self-care, productivity, and leisure activities. The caregiver is asked to identify the activities that is needed and difficult to be completed by their children. The importance of the five most necessary and difficult activities are scored by each caregiver on a ten-point scoring scale. The performance and satisfaction of the five most necessary, difficult and important activities are scored by each client and caregiver on a 10-point scale. The scores of performance or satisfaction scale were aggregated on the five most necessary, difficult and important activities.

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Jiun Shie, Dr., Principal Investigator — National Pingtung University
Locations (2):
- Taiwan (2):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City